CLINICAL TRIAL: NCT05383833
Title: Creatine to Augment Bioenergetics in Alzheimer's
Acronym: CABA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Collaborators: Alzheimer's Association (Other)
Responsible Party: Principal Investigator, Matthew Taylor, Assistant Professor, University of Kansas Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 148507
Record Dates: First submitted 2022-04-20; First posted 2022-05-20 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-08

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Creatine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Creatine Monohydrate Arm (Experimental): This study a single arm intervention. All participants will receive 20 grams of creatine monohydrate daily for the whole intervention (8 weeks).
  Interventions: Dietary Supplement: Creatine Monohydrate

INTERVENTIONS:
Dietary Supplement: Creatine Monohydrate — Participants will take 20 grams of creatine monohydrate daily for 8 weeks.The 20 grams will be divided into two equal 10 gram doses that will be stirred into a beverage. One 10 gram dose will be taken in the morning and the other 10 gram dose in evening.

SUMMARY:
By doing this study, researchers hope to see if creatine monohydrate is a helpful treatment for people with Alzheimer's disease.

DETAILED DESCRIPTION:
Alzheimer's disease is a progressive brain disorder that causes memory and thinking problems. Current medications may temporarily help with symptoms but cannot stop the disease from getting worse. As such, new treatments that slow or stop the disease from progressing are needed.

There is some evidence from animal studies that taking creatine monohydrate may improve thinking in Alzheimer's disease and be good for brain health. However, no studies have looked at creatine monohydrate supplementation in humans with Alzheimer's.

Creatine monohydrate is a dietary supplement regulated by the FDA. This is a study that will test if taking creatine monohydrate may be a helpful treatment for people with Alzheimer's disease. In this study, investigators will will evaluate:

1. Whether persons with Alzheimer's disease are able to easily take creatine monohydrate for 8 weeks.
2. Whether creatine monohydrate affects thinking function in people with Alzheimer's Disease.
3. Whether creatine monohydrate affects certain biochemicals in the brain and body.
4. Whether creatine monohydrate improves muscle size and strength.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed cognitive impairment due to Alzheimer's disease
* Agreed cooperation from a study partner
* Speaks English as primary language
* Age 60 to 90
* Stable medication for ≥30 days
* BMI ≥ 20.0kg/m2

Exclusion Criteria:

* Insulin-requiring diabetes, cancer requiring chemotherapy or radiation within the past 5 years, or recent cardiac event (i.e., heart attack, etc.)
* Other neurodegenerative disease
* Ongoing renal disorder or abnormal renal or liver function
* Unable to undergo MRI
* Clinical trial or investigational drug or therapy participation within 30 days of the screening visit
* Non-English speakers
* Inability to perform strength testing
* Weight > 350 lbs.

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-12-12 (Actual); Primary Completion 2024-05-14 (Actual); Study Completion 2024-05-14 (Actual)

PRIMARY OUTCOMES:
Adherence to Creatine Monohydrate Intervention | 8 weeks
  Participants will keep a daily supplement tracker (with the help of a consenting study partner). They will also bring unconsumed creatine monohydrate powder to study visits where study personnel will measure and validate against expected intake.
Change in Blood Creatine | Baseline, 4 weeks, and 8 weeks
  Measure of serum creatine levels at baseline, 4 weeks, and 8 weeks.

SECONDARY OUTCOMES:
Change in Brain Creatine Status | Baseline and 8 weeks
  Brain total creatine levels are measured in the brain using magnetic resonance spectroscopy in a 3 T clinical scanner.
Change in Cognition | Baseline and 8 weeks
  NIH Toolbox (NIH-TB) Cognition Battery will be used to assess changes in a composite global cognition score at baseline and 8 weeks.
Change in Peripheral Mitochondrial Respiration | Baseline and 8 weeks
  Blood platelet and leukocyte mitochondrial respiration (oxygen consumption) will be determined using the Oroboros Oxygraph-2K system.
Change in Muscle Strength | Baseline and 8 weeks
  Muscle strength will be tested on the right quadriceps femoris (upper leg) using an isokinetic dynamometer.
Change in Muscle Size | Baseline and 8 Weeks
  Muscle size of the right quadriceps femoris (upper leg) will be determined using ultrasonography (ultrasound).

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Taylor, PhD, RD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Smith AN, Sullivan DK, Morris JK, Carbuhn AF, Herda TJ, Taylor MK. Eight weeks of creatine monohydrate supplementation is associated with increased muscle strength and size in Alzheimer's disease: data from a single-arm pilot study. Front Nutr. 2025 Sep 4;12:1670641. doi: 10.3389/fnut.2025.1670641. eCollection 2025. PMID 40977987
- [Derived] Smith AN, Choi IY, Lee P, Sullivan DK, Burns JM, Swerdlow RH, Kelly E, Taylor MK. Creatine monohydrate pilot in Alzheimer's: Feasibility, brain creatine, and cognition. Alzheimers Dement (N Y). 2025 May 19;11(2):e70101. doi: 10.1002/trc2.70101. eCollection 2025 Apr-Jun. PMID 40395689
- [Derived] Taylor MK, Burns JM, Choi IY, Herda TJ, Lee P, Smith AN, Sullivan DK, Swerdlow RH, Wilkins HM. Protocol for a single-arm, pilot trial of creatine monohydrate supplementation in patients with Alzheimer's disease. Pilot Feasibility Stud. 2024 Feb 27;10(1):42. doi: 10.1186/s40814-024-01469-5. PMID 38414003